CLINICAL TRIAL: NCT02616783
Title: A Phase 3b, Randomized, Open-Label Study to Evaluate Switching From a Tenofovir Disoproxil Fumarate (TDF) Containing Regimen to Elvitegravir/Cobicistat/Emtricitabine/ Tenofovir Alafenamide (E/C/F/TAF) Fixed-Dose Combination (FDC) in Virologically-Suppressed, HIV-1 Infected Subjects Aged ≥ 60 Years
Brief Title: Switching From a Tenofovir Disoproxil Fumarate (TDF) Containing Regimen to Elvitegravir/Cobicistat/Emtricitabine/ Tenofovir Alafenamide (E/C/F/TAF) Fixed-Dose Combination (FDC) in Virologically-Suppressed, HIV-1 Infected Adults Aged ≥ 60 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-292-1826; 2015-002712-32 (EudraCT Number)
Record Dates: First submitted 2015-11-23; First posted 2015-11-30 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2019-01

CONDITIONS: HIV-1 Infection
Keywords: HIV 1 Infection; HIV; Virologically-Suppressed
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- E/C/F/TAF (Experimental): Participants will switch from tenofovir disoproxil fumarate (TDF) and emtricitabine (FTC) or 3TC plus a third agent to E/C/F/TAF and will receive treatment for 48 weeks.
  Interventions: Drug: E/C/F/TAF
- Remain current regimen (Active Comparator): Participants will remain on current TDF and FTC (or FTC/TDF) or 3TC plus continuing third agent.
  Interventions: Drug: TDF; Drug: FTC; Drug: FTC/TDF; Drug: 3TC; Drug: Third agent

INTERVENTIONS:
Drug: E/C/F/TAF — 150/150/200/10 mg FDC tablet administered orally once daily
  Other Names: Genvoya®
  Arms: E/C/F/TAF
Drug: TDF — 300 mg tablet administered orally once daily
  Other Names: Viread®
  Arms: Remain current regimen
Drug: FTC — 200 mg capsule administered orally once daily
  Other Names: Emtriva®
  Arms: Remain current regimen
Drug: FTC/TDF — 200/300 mg tablet administered orally once daily
  Other Names: Truvada®
  Arms: Remain current regimen
Drug: 3TC — Tablet administered orally
  Other Names: Lamivudine; Epivir®
  Arms: Remain current regimen
Drug: Third agent — Third agent may include one of the following regimens: lopinavir+ritonavir (LPV/r; Kaletra®), atazanavir (ATV; Reyataz®) + ritonavir (RTV; Norvir®), ATV + cobicistat (COBI;Tybost®) (or ATV/COBI FDC), DRV + RTV, darunavir (DRV; Prezista®) + COBI (or DRV/COBI FDC), fosamprenavir (FPV; Lexiva®) + RTV , saquinavir (SQV; Invirase®; Fortovase®) + RTV, efavirenz (EFV;Sustiva®), rilpivirine (RPV;Edurant®), nevirapine (NVP;Viramune®), etravirine (ETR;Intelence®), raltegravir (RAL; Isentress®), elvitegravir (EVG) + COBI, or dolutegravir (DTG;Tivicay®)
  Drug classes:
  * Protease inhibitors (PI): LPV/r, ATV, RTV, ATV, DRV, FPV, and SQV
  * Pharmacokinetic enhancer: COBI
  * Non-nucleoside reverse transcriptase inhibitors (NNRTI): EFV, RPV, NVP, and ETR
  * Integrase inhibitors: RAL and DTG
  Arms: Remain current regimen

SUMMARY:
The primary objective of this study is to evaluate the safety of elvitegravir/cobicistat/emtricitabine/ tenofovir alafenamide (E/C/F/TAF) relative to unchanged current antiretroviral therapy (ART) by assessing spine and hip bone mineral density (BMD) measured at Week 48 in virologically-suppressed, HIV-1 infected participants aged ≥ 60 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Currently receiving a TDF and FTC or 3TC-containing 'backbone' (maximum 2 NRTIs) regimen plus a third agent for ≥ 6 consecutive months prior to screening visit. For individuals with 3 or more ART regimens, a regimen history must be provided for approval by the Sponsor.

Refer to assigned interventions for allowed third agents of the current regimen.

* Documented plasma HIV-1 RNA levels < 50 copies/mL for ≥ 6 months preceding the screening visit (measured at least twice using the same assay). In the preceding 6 months prior to screening, one episode of "blip" (HIV-1 RNA > 50 and < 400 copies/mL) is acceptable, only if HIV-1 RNA is < 50 copies/mL immediately before and after the "blip".
* Plasma HIV-1 RNA level < 50 copies/mL at screening visit
* Adequate renal function
* Estimated glomerular filtration rate ≥ 30 mL/min according to the Cockcroft-Gault formula (eGFRCG) and are on ARVs that are appropriately dose adjusted for renal function per package insert
* All documented historical plasma genotype(s) must not show resistance to TDF or FTC, including, but not limited to the presence of reverse transcriptase resistance mutations K65R, K70E, M184V/I, or thymidine analog-associated mutations (TAMs) that include M41L, L210W, D67N, K70R, T215Y/F, K219Q/E/N/R. If historical plasma prior to first ART is not available or individual has 3 or more ART regimens, individuals will have proviral genotype analysis prior to Day 1 to confirm absence of archived resistance to TDF or FTC.
* Study performed dual energy x-ray absorptiometry (DXA) scan and T-score received prior to Day 1

Key Exclusion Criteria:

* Previous use of any approved or experimental integrase strand transfer inhibitor (INSTI) (for any length of time) if the current regimen contains a PI/r
* Individuals will have no evidence of previous virologic failure on a PI/r or INSTI-based regimen (with or without resistance to either class of ARV)
* A new AIDS-defining condition diagnosed within the 30 days prior to screening (except CD4+ cell count and/or percentage criteria)
* Hepatitis C virus that would require therapy during the study
* Individuals receiving ongoing treatment for bone disease (eg, osteoporosis), including bisphosphonates, denosumab, and strontium ranelate

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (35):
- Belgium (2):
  - CHU Saint-Pierre University Hospital, Brussels
  - University Hospital Gent, Ghent
- France (11):
  - CHU - Groupe Saint-Andre, Bordeaux
  - CHU de Dijon, Dijon
  - Hopital Europeen Marseille, Marseille
  - C.H.U. de Nantes, Nantes
  - C.H.U. de NICE, Nice
  - CHU Hotel Dieu, Paris
  - Hopital Necker les Enfants Malades, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Saint Louis, Paris
  - Hopital Haut-Leveque, Pessac
  - Service des Maladies Infectieuses et du Voyageur, Tourcoing
- Italy (9):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Busto Arsizio Hospital, Busto Arsizio
  - IRCCS A.O.U. San Martino, Genova
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Azienda Ospedaliero Universitaria Policlinico di Modena, Modena
  - U.O. Malattie Infettive, Pescara
  - Istituto Nazionale Malattie Infettive Lazzaro Spallanzani I.R.C.C.S., Roma
  - Azienda Ospedaliero Universitaria di Sassari, Sassari
  - Dipartimento di Malattie Infettive e Tropicali, Torino
- Spain (10):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Ramon Y Cajal University Hospital, Madrid
  - Hospital Costa Del Sol, Marbella
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (3):
  - Royal Victoria Hospital, Belfast
  - Mortimer Market Centre, London
  - Newcastle Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Derived] Maggiolo F, Rizzardini G, Raffi F, Pulido F, Mateo-Garcia MG, Molina JM, Ong E, Shao Y, Piontkowsky D, Das M, McNicholl I, Haubrich R. Bone mineral density in virologically suppressed people aged 60 years or older with HIV-1 switching from a regimen containing tenofovir disoproxil fumarate to an elvitegravir, cobicistat, emtricitabine, and tenofovir alafenamide single-tablet regimen: a multicentre, open-label, phase 3b, randomised trial. Lancet HIV. 2019 Oct;6(10):e655-e666. doi: 10.1016/S2352-3018(19)30195-X. PMID 31578954

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe. The first participant was screened on 22 December 2015. The last study visit occurred on 21 March 2018.
Pre-assignment Details: 214 participants were screened.
Groups:
- E/C/F/TAF: Participants switched from tenofovir disoproxil fumarate (TDF) and emtricitabine (FTC) or 3TC plus a third agent to elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) (150/150/200/10 mg) fixed-dose combination (FDC) tablet once daily for 48 weeks.
- Stay on Baseline Regimen: Participants stayed on current regimen of TDF and FTC (or FTC/TDF) or 3TC plus continuing third agent for 48 weeks.
Period: Overall Study
Arm/Group | E/C/F/TAF | Stay on Baseline Regimen
Started | 111 | 56
Completed | 105 | 54
Not Completed | 6 | 2
Not completed — Randomized but Not Treated | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0
Not completed — Non-Compliance with Study Drug | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrew Consent | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were randomized into the study and received at least 1 dose of study drug.
Groups:
- E/C/F/TAF: Participants switched from TDF and FTC or 3TC plus a third agent to E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | E/C/F/TAF | Stay on Baseline Regimen | Total
Number analyzed (Participants) | 110 | 56 | 166
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65 (4.6) | 66 (4.9) | 66 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 96 | 51 | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 8 | 24
  Not Hispanic or Latino | 88 | 42 | 130
  Unknown or Not Reported | 6 | 6 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 103 | 49 | 152
  Not Permitted | 5 | 4 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 8 | 1 | 9
  Italy | 36 | 15 | 51
  United Kingdom | 8 | 3 | 11
  France | 29 | 23 | 52
  Spain | 29 | 14 | 43
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 109 | 56 | 165
  ≥ 50 copies/mL | 1 | 0 | 1
CD4+ Cell Count [Mean (Standard Deviation); unit: cells/µL] | 649 (255.6) | 676 (316.5) | 658 (277.0)
CD4+ Cell Count Category [Count of Participants; unit: Participants]
  ≥ 50 to < 200 cells/µL | 0 | 2 | 2
  ≥ 200 to < 350 cells/µL | 12 | 8 | 20
  ≥ 350 to < 500 cells/µL | 18 | 7 | 25
  ≥ 500 cells/µL | 80 | 39 | 119
Spine Bone Mineral Density (BMD) [Mean (Standard Deviation); unit: g/cm^2] — Population: The Spine Dual-Energy X-ray Absorptiometry (DXA) Analysis Set included all participants who were randomized into the study, received at least 1 dose of study drug, had non missing screening spine BMD values, and did not have any major protocol violations.
  g/cm^2
    number analyzed (Participants) | 109 | 55 | 164
    (all) | 1.036 (0.1886) | 1.052 (0.1789) | 1.042 (0.1850)
Hip BMD [Mean (Standard Deviation); unit: g/cm^2] — Population: The Hip DXA Analysis Set included all participants who were randomized into the study, received at least 1 dose of study drug, had non missing screening hip BMD values, and did not have any major protocol violations.
  g/cm^2
    number analyzed (Participants) | 109 | 55 | 164
    (all) | 0.922 (0.1332) | 0.927 (0.1346) | 0.924 (0.1332)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 48 in Spine BMD
Time Frame: Baseline; Week 48
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | E/C/F/TAF | Stay on Baseline Regimen
Number analyzed (Participants) | 102 | 54
Percent change | 2.237 (3.2727) | -0.104 (3.3854)
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Regimen; Test type: Superiority; p < 0.001, ANOVA; P-value was calculated using the ANOVA model with baseline spine BMD score, sex, and treatment as fixed effects; Difference in Percentages = 2.427, 95% CI 2-sided [1.337 to 3.517] — The 95% confidence intervals (CI) were calculated using the ANOVA model with baseline spine BMD score, sex, and treatment as fixed effects

2. Primary Outcome: Percent Change From Baseline to Week 48 in Hip BMD
Time Frame: Baseline; Week 48
Population: Participants in the Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | E/C/F/TAF | Stay on Baseline Regimen
Number analyzed (Participants) | 101 | 54
Percent change | 1.330 (2.1968) | -0.726 (3.2069)
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Regimen; Test type: Superiority; p < 0.001, ANOVA; P-value was calculated using the ANOVA model with baseline hip BMD score, sex, and treatment as fixed effects; Difference in percentages = 2.036, 95% CI 2-sided [1.168 to 2.904] — The 95% CIs were calculated using the ANOVA model with baseline hip BMD score, sex, and treatment as fixed effects

3. Secondary Outcome: Percent Change From Baseline to Week 24 in Spine BMD
Time Frame: Baseline; Week 24
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | E/C/F/TAF | Stay on Baseline Regimen
Number analyzed (Participants) | 104 | 54
Percent change | 1.625 (3.2346) | -0.027 (2.9875)
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Regimen; Test type: Superiority; p < 0.001, ANOVA; P-value was calculated using the ANOVA model with baseline spine BMD score, sex, and treatment as fixed effects; Difference in percentages = 1.749, 95% CI 2-sided [0.726 to 2.771] — The 95% CIs were calculated using the ANOVA model with baseline spine BMD score, sex, and treatment as fixed effects

4. Secondary Outcome: Percent Change From Baseline to Week 24 in Hip BMD
Time Frame: Baseline; Week 24
Population: Participants in the Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | E/C/F/TAF | Stay on Baseline Regimen
Number analyzed (Participants) | 103 | 54
Percent change | 0.808 (1.9084) | -0.537 (2.7647)
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Regimen; Test type: Superiority; p < 0.001, ANOVA; P-value was calculated using the ANOVA model with baseline hip BMD score, sex, and treatment as fixed effects; Difference in percentages = 1.351, 95% CI 2-sided [0.602 to 2.099] — The 95% CIs were calculated using the ANOVA model with baseline hip BMD score, sex, and treatment as fixed effects

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Full Analysis Set included all participants who were randomized into the study, received at least 1 dose of study drug, and did not have any major protocol violations.
Measure: Number; unit: Percentage of participants
Arm/Group | E/C/F/TAF | Stay on Baseline Regimen
Number analyzed (Participants) | 109 | 55
Percentage of participants | 94.5 | 100.0
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Regimen; Test type: Superiority; p = 0.18, Fisher Exact — P-values for the superiority test comparing the percentages of participants with HIV-1 RNA < 50 copies/mL were from the Fisher exact test; Difference in percentages = -5.5, 95% CI 2-sided [-11.8 to 1.6] — Differences in percentages and 95% CI were generated based on exact method

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | E/C/F/TAF | Stay on Baseline Regimen
Number analyzed (Participants) | 109 | 55
Percentage of participants | 93.6 | 94.5
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Regimen; Test type: Superiority; p = 1.00, Fisher Exact; P-values for the superiority test comparing the percentages of participants with HIV-1 RNA < 50 copies/mL were from the Fisher exact test; Difference in percentages = -1.0, 95% CI 2-sided [-8.5 to 9.3] — Differences in percentages and 95% CI were generated based on exact method

7. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | E/C/F/TAF | Stay on Baseline Regimen
Number analyzed (Participants) | 99 | 54
cells/μL | 48 (161.9) | -4 (153.9)
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Regimen; Test type: Superiority; p = 0.053, ANOVA; The p-value, difference in least square means (LSM), and its 95% CI were from ANOVA model with treatment as a fixed effect; Difference in LSM = 52, 95% CI 2-sided [-1 to 106]

8. Secondary Outcome: Change in Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | E/C/F/TAF | Stay on Baseline Regimen
Number analyzed (Participants) | 102 | 50
cells/μL | 56 (177.7) | -1 (149.1)
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Regimen; Test type: Superiority; p = 0.051, ANOVA; The p-value, difference in LSM, and its 95% CI were from ANOVA model with treatment as a fixed effect; Difference in LSM = 57, 95% CI 2-sided [0 to 115]

ADVERSE EVENTS:
Time Frame: Up to 48 weeks plus 30 days
Description: Safety Analysis Set included participants who were randomized into the study and received at least 1 dose of study drug.
Arm/Group | E/C/F/TAF | Stay on Baseline Regimen
All-Cause Mortality (participants affected / at risk) | 1/110 | 0/56
Serious Adverse Events (participants affected / at risk) | 10/110 | 1/56
Other Adverse Events (participants affected / at risk) | 47/110 | 20/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF (N=110) | Stay on Baseline Regimen (N=56)
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Neuritis cranial (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF (N=110) | Stay on Baseline Regimen (N=56)
Diarrhoea (Gastrointestinal disorders) | 8 | 2
Bronchitis (Infections and infestations) | 4 | 6
Nasopharyngitis (Infections and infestations) | 12 | 3
Urinary tract infection (Infections and infestations) | 4 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Hypertension (Vascular disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol: Original (2015-07-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT02616783/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT02616783/Prot_001.pdf
  • Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT02616783/SAP_002.pdf